CLINICAL TRIAL: NCT01518751
Title: Orthostatic Dysregulation and Associated Gastrointestinal Dysfunction in Parkinson's Disease - Evolution A Monocentric Study to Investigate the Development of Symptoms of Autonomic Dysregulation in Parkinson's Disease
Brief Title: Orthostatic Dysregulation and Associated Gastrointestinal Dysfunction in Parkinson's Disease - Evolution
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-NR. 2011-0077
Record Dates: First submitted 2012-01-17; First posted 2012-01-26 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Parkinson's Disease - Autonomic Dysregulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Symptoms of blood pressure dysregulation, impaired swallowing and digestion are common amongst parkinson patients. The overall aim of this study is to examine blood pressure regulation and esophageal motility and gastric emptying in Parkinson's disease (PD) patients.

The investigators hypothesize that - compared to age-matched controls - PD patients display an altered regulation of blood pressure, altered gastroesophageal motility, and delayed gastric emptying. These symptoms occur already early in the disease process, but aggravate with progression of the disease.

The investigators will perform a 7-day blood pressure measurement, measurement of central blood pressure and pulse wave velocity, assessment of pulse variability, Schellong tests to assess orthostatic function, high resolution manometry assessments during swallowing acts, and a 13C-sodium octanoate breath test to assess gastric emptying, in 18 PD patients (9 each Hoehn&Yahr stages 1,2) and 12 age- and gender-matched healthy controls. Results will be interpreted in relation to the severity of PD motor symptoms.

The investigators anticipate that blood pressure dysregulation and gastroesophageal motility disturbances will be present only in PD subjects, but not in matched controls without neurological disorders and without any extrapyramidal motor signs. Furthermore, the investigators expect to find an association between motor impairment and the severity of these autonomic symptoms, however, that according to the Braak staging, subtle disturbances must already be present in the early stages of PD.

ELIGIBILITY:
Inclusion criteria: - informed, written & formal consent for participation

* male/female subjects, aged 50-70 years
* PD patients (9 subjects each in Hoehn & Yahr stage 1 & 2)

Exclusion criteria: - Antihypertensive treatment

* medication influencing gastrointestinal motility for at least the elimination half life of the drug
* medication interfering with blood-pressure regulation for at least the elimination half life of the drug
* significant systemic illness
* BMI < 18 or > 30kg/m2
* symptoms or a history of GI disease or surgery
* with any evidence of infectious disease
* evidence or history of drug or alcohol abuse
* diabetes mellitus

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects included in this trial must fulfil the he following criteria:
  * informed, written & formal consent for participation
  * male / female subjects, aged 50-70 years
    18 PD patients
  * 9 subjects Hoehn & Yahr stage 1, disease duration <4 years
  * 9 subjects Hoehn & Yahr stage 2; disease duration 4-8 years
    12 healthy control subjects
  * age- and gender-matched
  * without signs or history of neurological disorders
  * without significant systemic comorbidities (malignant / cardiovascular)
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
orthostatic hypotension | during study visit
  drop of systolic (≥20mmHg) or diastolic (≥10mmHg) blood pressure upon Schellong test

SECONDARY OUTCOMES:
delayed gastric emptying | during study visit
  statistical difference in mean gastric emptying assessed via octanoate breath test
long term blood pressure | during 7d after study visit at home
  mean 7d systolic, diastolic, mean arterial blood pressure and heart rate recordings
heart rate variability | during study visit
  difference in heart rate variability or spectral analysis of heart rate variability?
arterial stiffening | during study visit
  difference in pulse wave velocity and augmentation index calculation from applanation tonometry recordings?
oesophageal motility | during study visit
  high-density manometry to measure aspects of oesophageal motility
subjective symptoms of gastrointestinal and cardiovascular dysfunction | during study visit
  validated questionnaires: Fraser, 2007, p14133; Stanghellini, 1996, p14183; Revicki, 2003, p13823; Kaufmann, 2012, p13817; }
Clinical assessment | during study visit
  UPDRS part III and MoCA score (Nasreddine, 2005, p14186)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Baumann, Ass. Prof., MD, Principal Investigator — University Hospital Zurich, Neurology
Locations (1):
- University Hospital Zurich, Neurology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Epprecht L, Schreglmann SR, Goetze O, Woitalla D, Baumann CR, Waldvogel D. Unchanged gastric emptying and visceral perception in early Parkinson's disease after a high caloric test meal. J Neurol. 2015 Aug;262(8):1946-53. doi: 10.1007/s00415-015-7799-z. Epub 2015 Jun 6. PMID 26048686